CLINICAL TRIAL: NCT03277885
Title: Evaluation of the Prevalence of Pain Disorders in a Professional Context Among Employees of French Furniture Shop.
Brief Title: Prevalence of Pain Disorders in Employees of French Furniture Shop.
Acronym: PREVADouleur
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-347
Record Dates: First submitted 2017-09-04; First posted 2017-09-11 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Chronic Pain
Keywords: Work related chronic pain; Preventive care
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: chronic pain — work related chronic pain

SUMMARY:
In France, the Direction of Research, Studies, Evaluation and Statistics, in their 2015 report on "Chronic pain: the state of health of the population in France - Indicators associated with the Public health ", shows that 34.6% of the working population declare themselves to be facing psycho-social risks, including chronic pain disorders.

The main survey conducted in France on chronic pain showed that 32% of French people expressed daily pain for more than 3 months, with 20% reporting chronic pain of moderate or severe intensity. According to a report by the HAS in 2009, about 30% of patients consulting for pain in pain center (CETD) are working and 20% are on sick leave or work-related accidents.

Chronic pain would also be responsible in France for the limitation of professional activities in 6% of 25-64 year olds, 15% job losses, 12% changes in work responsibilities, 12% changes in employment and 18 % of associated depressions. In addition, 40% of chronic pain patients experienced a direct impact at work: loss, change in responsibilities and activity.

Combined with the difficulty of understanding and thus treating chronic pain, these data demonstrate the challenge faced by occupational health services in their preventive, curative and palliative approach to chronic pathologies. Innovation for any new prevention and therapy for chronic pain then becomes necessary.

The main objective of this first study will be the evaluation of the prevalence of pain disorders among the employees of French furniture shop. .

DETAILED DESCRIPTION:
In order to have the earliest possible representativeness of French furniture shop, a "virtual" store will be created from 400 volunteer employees from 14 French furniture shop. Each job will be represented and the number of employees per job will respect the average proportion observed in the French furniture shop.

Following the on-site presentation of the details of the survey, by a doctor from Clermont-Ferrand University Hospital, volunteers will be informed within their company of the start of the survey. Each volunteer employee will have access to the information document (paper format) explaining in detail the purpose, content and conduct of the survey. If the voluntary collaborator agrees to participate, he / she will be asked to respond to the survey via the computer platform of the Clermont-Ferrand University Hospital.

Before completing the questionnaires, the employee will be asked to participate in the survey, via a YES / NO choice on the computer platform, which will serve as proof of non-opposition. The employee will be free to reverse his initial decision at any time by informing the coordinating center.

Volunteers who have agreed to participate in the study will be asked to respond to the survey questionnaires during each survey. Volunteers will have no obligation to participate in all investigations.

The data manager of the coordinating center will build a specific and secure platform via the REDCap website (http://project-redcap.org/). Volunteer collaborators will be provided with the web link to respond to the survey directly on the REDCap platform at their workplace or at home.

The deployment of the survey to employees will be carried out over a period of 1 month.

This survey will take place in 4 separate campaigns with a 4-month interval: October / February / June / October (to give an overview of the season effect on the data, as well as a longitudinal aspect). During each campaign, employees will be notified and can participate in the survey. Each employee may participate in one or more investigations.

ELIGIBILITY:
Inclusion Criteria:

* All voluntary employees of French furniture shop
* Non-opposition to participation in the study

Exclusion Criteria:

* Employees unable to understand or answer questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: employees of French furniture shop
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of painful disorders | At the end of each survey campaign (a campaign lasts 1 month and is repeated every 4 months for 12 months, a total of 4 campaigns).
  An employee will be considered painful if the pain intensity is greater than 3/10 on a numerical rating scale (0 = no pain at 10 = worst possible pain).

SECONDARY OUTCOMES:
Sociodemographic characterization | at day 1
  Questionnaires
Number of medical and paramedical visits over the past 12 months for a cause of pain. | during each survey campaign (4 campaigns over a 12-month period).
  Questionnaires
Anxiety and Depression Score | at day 1
  Questionnaire HADS
Quality of life | at day 1
  Questionnaire SF-12
Catastrophism | at day 1
  Questionnaire PCS
Characterization of pain | at day 1
  Questionnaire BPI
Characterization of kinesiophobia | at day 1
  Questionnaire TSK
Screening for neuropathic pain | at day 1
  Questionnaire DN4 interview
Characterization of lumbar pain. | at day 1
  Questionnaire FABQ

CONTACTS AND LOCATIONS:
Overall Officials: Christian DUALE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France